CLINICAL TRIAL: NCT02904889
Title: Stimulating Engagement in Daily and Physical Activities Among Older Adults Receiving Homecare Services: An Exploratory Trial (Part of Basic Care Revisited)
Brief Title: Stimulating Engagement in Daily and Physical Activities Among Older Adults Receiving Homecare Services (Part of Basic Care Revisited)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Silke Metzelthin, PhD, Maastricht University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZonMw no. 520002003
Record Dates: First submitted 2016-09-08; First posted 2016-09-19 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2016-12

CONDITIONS: Community-dwelling Older Adults

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stay Active at Home (Experimental): One group of homecare professionals receives a training programme. In this training they learn to motivate their clients to be more active in daily and physical activities.
  Interventions: Behavioral: Stay Active at Home
- Usual care (Active Comparator): Second group of homecare professionals will get no training and their clients will receive usual homecare.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Stay Active at Home — Stay Active at Home' aims to change the behaviour of community nurses and domestic support workers by offering them an intensive training programme. Subsequently, professionals are expected to deliver goal-oriented, holistic and person-centred services focusing on supporting older adults to maintain, gain or restore their competences to engage in physical and daily activities so that they can manage their everyday life as independently as possible.
  Arms: Stay Active at Home
Other: Usual care — Homecare professionals will get no training and their clients will receive usual homecare.
  Arms: Usual care

SUMMARY:
Most older adults want to stay at home for as long as possible. To reach this aim it is important to maintain their mobility and self-care abilities. However, many older adults are at risk to lose their abilities, as they have an inactive lifestyle. In this study, homecare professionals learn to motivate their clients to be more active in daily and physical activities. Examples of these activities are washing and dressing, household chores or going for a walk.

The primary aim of this exploratory study is to evaluate the implementation of the 'Stay Active at Home' program (process evaluation). The secondary aim is to get insight into the potential effectiveness of the program with regard to several primary and secondary outcomes measures (effect evaluation). The tertiary aim is to test the feasibility of the proposed study design.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years
* Community-dwelling
* Indication for homecare
* ≥10 hours sedentary behaviour/day (measured with LASA vragenlijst questionnaire)
* Written informed consent

Exclusion Criteria:

* Terminal
* Serious cognitive or psychological problems
* Not able to speak Dutch

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (older adults) | after 6 months
Groningen Activity Restriction Scale (older adults) | after 6 months

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (older adults) | baseline, after 6 and 9 months
EQ-5D-5L (older adults) | baseline, after 6 and 9 months
Healthcare utilisation questionnaire (older adults) | baseline, after 6 and 9 months
Self-efficacy and outcome expectation questionnaire (older adults and professionals) | baseline, after 6 and 9 months
Satisfaction with care, 1 item CQ index (older adults) | baseline, after 6 and 9 months
Falls, 1 item 'How often did you fall during the ... months?' (older adults) | baseline, after 6 and 9 months
LASA sedentary behaviour questionnaire (older adults) | baseline, after 6 and 9 months
Physical activity (actigraph, counts/minute, subsample older adults) | baseline, after 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Gertrudis IJ Kempen, PhD, Study Chair — Maastricht University
Locations (1):
- MeanderGroep Zuid-Limburg, Kerkrade, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
data are avalailble upon request depending on specific circumstances